CLINICAL TRIAL: NCT04589065
Title: Pilot Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) to Treat Patients With NYHA Stage III or IV Heart Failure (HF) With Persistent Congestion and Worsening Renal Function as a Result of Cardiorenal Syndrome (CRS) That is Resistant to Optimal Medical Therapy Including Loop Diuretics
Brief Title: SCD for CRS in Congestive Heart Failure (CHF) (No Left Ventricular Assist Device)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment on hold pending amendment approval.
Sponsor: Lenar Yessayan (Other)
Responsible Party: Sponsor-Investigator, Lenar Yessayan, Professor of Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00178335
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Chronic Systolic Heart Failure; Renal Failure; Cardiorenal Syndrome
Keywords: Hospitalized
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Selective Cytopheretic Device (Experimental)
  Interventions: Device: Selective Cytopheretic Device

INTERVENTIONS:
Device: Selective Cytopheretic Device — SCD therapy will take place for 4 hours on day 1, 3, and 5 while on hemodialysis treatment. Participants will be continue to be followed until 30 days after the last SCD treatment.

SUMMARY:
The purpose of this clinical trial is to see if a new device (SCD) is safe and if it can reduce damage to the kidney enough to allow medications to work to improve heart and kidney function for use in patients that have moderate to severe heart failure and is at least in part due to heart failure and it not responding to standard medical therapy. The SCD is a cartridge used with a commercial hemodialysis unit.

Participants will be enrolled in the clinical trial once eligibility is confirmed. In addition to clinical assessments and laboratory testing participants will have surface echocardiograms during the trial. The SCD treatment will take place for 4 hours on day 1, 3, and 5 while on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Primary hospitalization for acute decompensated chronic systolic heart failure as defined:

  * Left ventricular ejection fraction ≤35% as confirmed by baseline imaging procedure.
  * New York Heart Association (NYHA) class III or IV chronic (≤ 90 days) systolic heart failure, with failure to respond to optimal medical therapy (beta blocker, Angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blockers (ARB) or valsartan/sacubitril, aldosterone antagonist, unless not tolerated or contraindicated, and loop diuretic, as needed) for 45 of the last 60 days.
* Baseline Estimated Glomerular Filtration Rate (eGFR)** ≥ 40 ml/min/1.73 m2 (baseline defined as the highest known eGFR within 90 days of study enrollment)
* Worsening renal failure (WRF), defined for the purposes of this study as increase serum creatinine ≥ 0.5 mg/dL from baseline (baseline defined as the lowest known serum creatinine within 90 days of study enrollment)
* Cardiorenal syndrome is the most likely explanation for WRF
* Persistent signs and /or symptoms of congestion (peripheral edema, dyspnea, pulmonary rales, neck vein distension) despite optimal medical therapy including intravenous diuretic therapy and an estimated need for greater than 5 kg. of fluid removal. For the purposes of this study, optimal intravenous diuretic therapy is defined as:

  * Furosemide equivalent total daily dose of 240 mg (furosemide 40mg=1mg bumetanide)
  * Furosemide equivalent dose given either as a single or multiple intravenous bolus or continuous infusion
  * A furosemide equivalent total daily dose <240 mg if the dose has resulted in >3000 ml urine output/24 hours

Exclusion Criteria:

* Prior sensitivity to dialysis device components
* Individual with known hypersensitivity to citrate
* Bacteremia or possible infection, as evidence by fever, white blood cell count > 10,000/microliter, or any other signs of acute or chronic infection, and any patient receiving antibiotic or antiviral therapy.
* Active malignancy requiring chemotherapy, biological therapy or radiation therapy.
* The use of intravenous iodinated contrast agent within the prior 72 hours or the anticipated use of such an agent during SCD therapy.
* Need for intravenous vasopressor (i.e., phenylephrine, vasopressin), intravenous. vasoconstricting inotrope (i.e., norepinephrine or epinephrine) or dopamine > 3 mcg/kg/min. (Note: use of vasodilating inotropes [i.e., dobutamine and milrinone] or dopamine at ≤ 3 mcg/kg/min will not preclude study inclusion).
* Persistent systolic blood pressure (SBP) < 80 mmHg.
* White blood cell (WBC)<4000/microliter.
* Platelets < 50,000/microliter.
* Serum creatinine > 4 mg/dL or receiving dialysis / continuous renal replacement therapy (CRRT)
* Acute coronary syndrome within the past month.
* Women who are pregnant, breastfeeding a child, or trying to become pregnant.
* Subject not able to sign informed consent.
* Use of any other investigational drug or device within the previous 30 days
* Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical studies where only measurements and/or samples are taken (i.e., no test device or test drug used) are allowed to participate.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cardiac Function - Left Ventricular Ejection Fraction | up to 4 weeks following last SCD treatment
  This will be assessed by surface echocardiography.

SECONDARY OUTCOMES:
Improved renal function as measured by serum creatinine | up to 4 weeks following the last SCD therapy
Improved renal function as measured by blood urea nitrogen (BUN) | up to 4 weeks following the last SCD therapy

CONTACTS AND LOCATIONS:
Overall Officials: Keith Aaronson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No